CLINICAL TRIAL: NCT01756183
Title: Exploratory Study on the S-1 + Paclitaxel Chemotherapy for Creating the Operation Chance in the Patients With Unresectable Gastric Cancer
Brief Title: Exploratory Study on the S-1 + Paclitaxel Chemotherapy for Unresectable Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPECIAL
Record Dates: First submitted 2012-11-29; First posted 2012-12-25 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: Surgically-Created Resection Cavity; Drug Safety
MeSH Terms: interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-1 + Paclitaxel Chemotherapy (Experimental): S-1: 60mg twice daily (after the breakfast and supper) for two weeks, and then suspend for one week.
  Paclitaxel: 150 mg/m2, iv, 3h, at D1
  Interventions: Drug: S-1 + Paclitaxel Chemotherapy

INTERVENTIONS:
Drug: S-1 + Paclitaxel Chemotherapy — Dose of S-1: 60mg bid，Twice daily (after the breakfast and supper) for two weeks, and then suspend for one week.
  Dose of Paclitaxel: 150 mg/m2, iv, 3h, at D1

SUMMARY:
Exploratory the S-1 + Paclitaxel Chemotherapy for Creating the Operation Chance in the Patients with Unresectable Gastric Cancer

DETAILED DESCRIPTION:
To assess the effectiveness and safety of S-1 + Paclitaxel for the peri-operative chemotherapy in Chinese patients with unresectable gastric cancer, so as to further find out the optimal protocol for the peri-operative chemotherapy in the patients with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

-Unresectable gastric cancer as proven histologically (AJCC, Version 7) under any following condition: Unable radical excision due to the local metastasis or invasion Metastasis to the lymph node beside the abdominal aorta Non-extensive metastasis to liver (not more than three metastatic foci of radical excision)

* Definitely diagnosed as above stage of stomach cancer before the operation via CT or MRI, ultrasonic endoscopy and blood tumor antigen test, or through the laparoscopy if necessary
* Untreated (e.g. radiotherapy, chemotherapy, target therapy and immunotherapy)
* ECOG (Eastern Cooperative Oncology Group) : 0~2
* Age: 18~75 years old
* Normal hemodynamic indices before the recruitment (including blood cell count and liver/kidney function). For example: WBC>4.0×109/L, NEU >1.5×109/L, PLT>100×109/L, BIL<1.5 times of upper limit of normal reference value, ALT and AST<2.5 times of upper limit of normal reference value, and CRE<1.2mg/dl
* Good cardiac function before the recruitment, no seizure of myocardial infarction in past half year, and controllable hypertension and other coronary heart diseases
* Not concomitant with other uncontrollable benign diseases before the recruitment (e.g. the infection in the lung, kidney and liver)
* Not participating in other study projects before and during the treatment
* Signed the Informed Consent Form

Exclusion Criteria:

* Not conforming to above inclusion criteria
* Distal metastasis to lung, brain and bone (except the liver)
* Ever operation on the stomach
* Operation intolerance due to other systemic basic diseases
* Ever administered other drugs (including TCM drugs) before the recruitment, or no guarantee of progress according to the study requirement after the recruitment
* Allergy to the drugs in this protocol
* Pregnant or lactating women
* Women at childbearing age and of pregnancy desire during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
radical resection rate | 3 months
  radical resection rate

SECONDARY OUTCOMES:
Adverse Events | 6 months
  Number and degree of Adverse Events
reaction rate | 2 months
  the reaction rate of chemotherapy
overall survival time | 3 years
  the overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: xiangdong Cheng, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China